CLINICAL TRIAL: NCT03815084
Title: Clinical Study on the Safety and Efficacy of PD1 Combined With DC-NK Cell in the Treatment of Solid Tumors
Brief Title: A Study of PD1 Combined With DC-NK Cell in the Treatment of Solid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Yunan Province/First People's Hospital of Yunan Provinve New Kunhua Hospital (Unknown); Henan Provincial People's Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PD-1/DC-NK YNYY-01
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — alpha-Synuclein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 and DC-NK treatment group (Experimental)
  Interventions: Drug: pd-1 and DC-NK cells

INTERVENTIONS:
Drug: pd-1 and DC-NK cells — total dose of 10ml KEYTRUDA® (pembrolizumab) will be administered at day0, 60million DC cells and 3 billion NK at day1, 3 billion NK cells at day2, 3 billion NK cells at day3 .

SUMMARY:
clinical study on the safety and efficacy of PD1 combined with dc-Nk in the treatment of solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Previously receiving ≥ first-line regimen chemotherapy;
2. Age over 3 years old and less than 14 years old;
3. The expected survival period is more than 3 months;
4. ECOG≤2;
5. Vital organ function is satisfied: cardiac ultrasound indicates cardiac ejection fraction ≥ 50%, no obvious abnormality in ECG; blood oxygen saturation ≥ 90%; creatinine clearance calculated by Cockcroft-Gault formula ≥ 40ml/min; ALT and AST ≤ 3 times the normal range, total bilirubin ≤ 2.0 mg / dl;
6. Blood routine: Hgb≥80g/L, ANC≥1×109/L, PLT≥50×109/L; There are measurable target lesions.

Exclusion Criteria:

1. Liver and kidney function:

   * Total bilirubin > 2 x ULN (Gilbert syndrome > 3 x ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 3 × ULN
   * Serum creatinine clearance >60mL/min
2. Serological examination:

   * Absolute neutrophil count (ANC) <0.75x109/L
   * Platelet count (PLT) <50x109/L
3. Active hepatitis B (HBV-DNA > 1000 copies / ml), hepatitis C, or uncontrolled infection;
4. The number of days of chemotherapy medication and the administration of hormones below 5mg is ≤3, and the number of days of withdrawal of hormones greater than 5mg is ≤5;
5. Active CNS disease (tumor cells in CSF);
6. Intracranial hypertension or unconsciousness; respiratory failure; diffuse vascular internal coagulation;
7. creatinine > 1.5 times the upper limit of normal or ALT / AST > 3 times the upper limit of normal or bilirubin > 2 times the upper limit of normal;
8. The New York Heart Association (NYHA) is classified as Level III or higher;
9. Uncontrolled diabetes;
10. With other uncontrolled diseases, the investigator believes that it is not suitable for joining;
11. Any situation that the investigator believes may increase the risk of the subject or interfere with the test results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
occurrence of treatment related adverse events | 1 year
  occurrence of treatment related adverse events that are possible, likely. Or definitely related to study treatment.

IPD SHARING:
Plan to Share IPD: No